CLINICAL TRIAL: NCT00110448
Title: Japanese Primary Prevention of Atherosclerosis With Aspirin for Diabetes (JPAD) Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kumamoto University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H14-Kouka(Seikatsu)-025
Record Dates: First submitted 2005-05-09; First posted 2005-05-10 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2008-08

CONDITIONS: Coronary Disease; Arteriosclerosis; Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; coronary heart diseases; primary prevention; atherosclerosis; aspirin
MeSH Terms: conditions — Coronary Disease; Arteriosclerosis; Diabetes Mellitus, Type 2; Atherosclerosis | interventions — Aspirin; N-acetyl-S-(alpha-methyl-4-(2-methylpropyl)benzeneacetyl)cysteine 4-(nitrooxy)butyl ester

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Aspirin use
  Interventions: Drug: Aspirin
- 2 (Active Comparator): No aspirin use
  Interventions: Drug: No aspirin

INTERVENTIONS:
Drug: Aspirin — Aspirin 81 mg or 100 mg per day
  Arms: 1
Drug: No aspirin — No aspirin use
  Arms: 2

SUMMARY:
The purpose of this study is to determine the effects of low-dose aspirin for the primary prevention of vascular events in patients with type 2 diabetes in Japan.

DETAILED DESCRIPTION:
There is a worldwide epidemic of diabetes and the number of individuals with diabetes is set to increase further. As individuals with diabetes are at high risk of accelerated atherosclerosis and thrombotic vascular events, the significant proportion of the cardiovascular disease burden is projected to be among this population. JPAD is a multicenter study with a prospective randomized open, blinded end-point (PROBE) design. The doses administered are aspirin 81 mg/day or 100 mg/day, the latter being enteric-coated Aspirin.

The primary objective was to compare the effect of aspirin on atherosclerotic events including cardiovascular events, cerebral vascular event, and other vascular events.

We also analyze hemorrhagic events in this RCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients have type 2 diabetes mellitus (30 or more years old and 85 years old or less).
* Patients give their informed consent to participate.

Exclusion Criteria:

* Patient has electrocardiographic changes, including ischemic ST-segment depression, ST-segment elevation, or pathologic Q waves.
* Patient has fixed ischemic heart disease, utilizing coronary angiography.
* Patient has cerebral vascular disease, including cerebral infarction, past hemorrhage, and experience of transient ischemic attack.
* Patient has arteriosclerotic disease, which needs internal medicine and/or surgical medical treatment.
* Patient has already taken the following anti-platelet or anti-thrombotic medicine: aspirin, ticlopidine, cilostazol, dipyridamole, trapidil, warfarin, and argatroban.
* Patient has severe gastric and/or duodenal ulcer.
* Patient has severe liver dysfunction.
* Patient has severe renal dysfunction.
* Patient has allergy for aspirin.
* Patient has atrial fibrillation.
* Pregnancy or the possible case of pregnancy.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2539 (Actual)
Dates: Start 2002-12; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Cardiovascular events | five years (median)
Cerebral vascular events | five years (median)
Aortic and peripheral vascular events, which needs internal medicine and/or surgical medical treatment | five years (median)

CONTACTS AND LOCATIONS:
Overall Officials: Hisao Ogawa, MD, Principal Investigator — Professor of Medicine, Department of Cardiovascular Medicine, Graduate School of Medical Sciences, Kumamoto University; Yoshihiko Saito, MD, Principal Investigator — Professor of Medicine, First Department of Internal Medicine, Nara Medical University
Locations (2):
- Japan (2):
  - Department of Cardiovascular Medicine, Graduate School of Medical Sciences, Kumamoto University, Kumamoto, Kumamoto
  - First Department of Internal Medicine, Nara Medical University, Kashihara, Nara

REFERENCES:
- [Derived] Matsumoto C, Ogawa H, Saito Y, Okada S, Soejima H, Sakuma M, Masuda I, Nakayama M, Doi N, Jinnouchi H, Waki M, Morimoto T. Incidence of atrial fibrillation in elderly patients with type 2 diabetes mellitus. BMJ Open Diabetes Res Care. 2022 Mar;10(2):e002745. doi: 10.1136/bmjdrc-2021-002745. PMID 35361621
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- [Derived] Matsumoto C, Ogawa H, Saito Y, Okada S, Soejima H, Sakuma M, Masuda I, Nakayama M, Doi N, Jinnouchi H, Waki M, Morimoto T; JPAD Trial Investigators; JPAD Trial Investigators:. Sex Difference in Effects of Low-Dose Aspirin on Prevention of Dementia in Patients With Type 2 Diabetes: A Long-term Follow-up Study of a Randomized Clinical Trial. Diabetes Care. 2020 Feb;43(2):314-320. doi: 10.2337/dc19-1188. Epub 2019 Dec 4. PMID 31801787
- [Derived] Saito Y, Okada S, Ogawa H, Soejima H, Sakuma M, Nakayama M, Doi N, Jinnouchi H, Waki M, Masuda I, Morimoto T; JPAD Trial Investigators. Low-Dose Aspirin for Primary Prevention of Cardiovascular Events in Patients With Type 2 Diabetes Mellitus: 10-Year Follow-Up of a Randomized Controlled Trial. Circulation. 2017 Feb 14;135(7):659-670. doi: 10.1161/CIRCULATIONAHA.116.025760. Epub 2016 Nov 15. PMID 27881565
- [Derived] Okada S, Morimoto T, Ogawa H, Kanauchi M, Nakayama M, Uemura S, Doi N, Jinnouchi H, Waki M, Soejima H, Sakuma M, Saito Y; Japanese Primary Prevention of Atherosclerosis With Aspirin for Diabetes Trial Investigators. Differential effect of low-dose aspirin for primary prevention of atherosclerotic events in diabetes management: a subanalysis of the JPAD trial. Diabetes Care. 2011 Jun;34(6):1277-83. doi: 10.2337/dc10-2451. Epub 2011 Apr 22. PMID 21515838
- [Derived] Saito Y, Morimoto T, Ogawa H, Nakayama M, Uemura S, Doi N, Jinnouchi H, Waki M, Soejima H, Sugiyama S, Okada S, Akai Y; Japanese Primary Prevention of Atherosclerosis With Aspirin for Diabetes Trial Investigators. Low-dose aspirin therapy in patients with type 2 diabetes and reduced glomerular filtration rate: subanalysis from the JPAD trial. Diabetes Care. 2011 Feb;34(2):280-5. doi: 10.2337/dc10-1615. PMID 21270185
- [Derived] Ogawa H, Nakayama M, Morimoto T, Uemura S, Kanauchi M, Doi N, Jinnouchi H, Sugiyama S, Saito Y; Japanese Primary Prevention of Atherosclerosis With Aspirin for Diabetes (JPAD) Trial Investigators. Low-dose aspirin for primary prevention of atherosclerotic events in patients with type 2 diabetes: a randomized controlled trial. JAMA. 2008 Nov 12;300(18):2134-41. doi: 10.1001/jama.2008.623. Epub 2008 Nov 9. PMID 18997198